#### **COVER PAGE**

**Official Title:** NON-INVASIVE NEURALLY ADJUSTED VENTILATORY ASSIST VERSUS NASAL INTERMITTENT POSITIVE PRESSURE VENTILATION FOR PRETERM INFANTS AFTER EXTUBATION: A RANDOMIZED CONTROLLED TRIAL

NCT number: NCT03388437

**Document Date:** 31/05/2021

# **Study Results**

| Study Type | Interventional |
|---|---|
| Study Design | Allocation: Randomized; Intervention Model: Parallel Assignment; Masking: None (Open Label); Primary Purpose: Treatment |
| Condition | Non-invasive neurally adjusted ventilatory assist versus nasal intermittent positive pressure ventilation for preterm infants after extubation |
| Intervention | Device: noninvasive respiratory support with <b>NAVA</b> mode and <b>NIPPV</b> |
| Enrollment | 36 |

# **Participant Flow**

| Recruitment Details | Patients recruited from single tertiary center neonatal intensive care | |
|---|---|---|
| | unit (NICU) level 3 at the King Fahad Armed Forces Hospital | |
| | in Saudi Arabia between May 2 | 2017 and April 2019 |
| <b>Pre-assignment Details</b> | 41 assessed for eligibility, 5 ex | xcluded, 36 randomized subsequently |
| | equally | |
| Arm/Group Title | NI-NAVA | NIPPV |
| Arm/Group Description | NI-NAVA after extubation | NIPPV after extubation |
| Arm/Group Description | Initial ventilatory settings | Positive Inspiratory Pressure (PIP) |
| | were NAVA level of 2; | incremented at 2 cm H2O from the |
| | Positive End Expiratory pre-extubation PEEP of 5-6 cm H2 | |
| | Pressure (PEEP) of 5-6 cm for 72 hours post extubation. The | |
| | H2O; apnea time 5-10 | respiratory rate was same as prior to |
| | seconds; and target electrical | extubation. |
| | activity of the diaphragm | |
| | (Edi) maximum between 10- | |
| | 15 and minimum <5 for 72 | |
| | hours post extubation. | |
| Period Title: Overall Stud | d Title: Overall Study | |
| Started | 18 | 18 |
| Completed | 18 | 18 |
| Not Completed | 0 | 0 |
| Reason Not Completed | | |
| Adverse Event (Death) | 2 | 1 |

## **Baseline Characteristics**

| Arm/C | Group Title | NI-NAVA<br>Group | NIPPV Group | Total |
|---|---|---|---|---|
| ▼ Arm/Group | Description | Non-invasive Neurally adjusted ventilatory assist (NAVA) after extubation in preterm infants | Non-invasive positive pressure ventilation (NIPPV) after extubation in preterm infants | Total of all reporting groups |
| Overall Number | of Baseline | 18 | 18 | 36 |
| <b>▼</b> Baseline Analysis Population Description | | [Not Specified] | | |
| Age at extubation, Continuous Mean (Standard deviation) Unit of measure: Days | | | | |
| | Number<br>Analyzed | 18 participants 1.67 (1.49) | 18 participants 1.17 (0.38) | 36<br>participants<br>1.41(1.11) |
| Sex: Female, Male | | | | |

| Measure Type: Count of Participants Unit of measure: Participants | | | | |
|---|---|---|---|---|
| | Number<br>Analyzed | 18 participants | 18 participants | 36 participants |
| | Female | 8 | 8 | 16 |
| | | 44.4% | 44.4% | 44.4% |
| | Male | 10 | 10 | 20 |
| | | 55.6% | 55.6% | 55.6%% |
| Gestational Age, | | | | |
| Mean (Standard<br>Deviation) | | | | |
| Unit of measure: Weeks | | | | |
| | Number<br>Analyzed | 18 participants | 18 participants | 36 participants |
| | | 28.94 (1.83) | 28.55 (1.18) | 28.74 (1.53) |
| Birth Weight, | | | | |
| Mean (Standard<br>deviation) | | | | |

| Unit of measure: g | | | | |
|---|---|---|---|---|
| | Number<br>Analyzed | 18 participants | 18 participants | 36 participants |
| | | 1251.94 (329.13) | 1051.0 (376.99) | 1151.47<br>(363.36) |
| Antenatal Steroid usage Measure Type: Count of Participants Unit of measure: Frequency | | | | |
| | Number<br>Analyzed | 18 participants | 18 participants | 36 participants |
| | YES | 14 (77.8%) | 11 (61.1%) | 25 (69.4%) |
| Presence of IUGR Measure Type: Count of Participants Unit of measure: Frequency | | | | |
| | Number<br>Analyzed | 18 participants | 18 participants | 36 participants |
| | | 0 (0%) | 1 (5.6%) | 1 (2.8%) |
| CRIB Score | | | | |

| Mean (Standard Deviation) Unit of measure: number | | | | |
|---|---|---|---|---|
| | Number<br>Analyzed | 18 participants | 18 participants | 36 participants |
| | | 1.72 (2.02) | 1.88 (1.40) | 1.80 (1.72) |
| Duration of invasive ventilation Mean (Standard Deviation) Unit of measure: hours | | | | |
| | Number<br>Analyzed | 18 participants | 18 participants | 36 participants |
| | | 22.77 (35.05) | 10.22 (11.55) | 16.50 (26.49) |
| Caffeine usage Measure Type: Count of Participants Unit of measure: Participants | | | | |
| | Number<br>Analyzed | 18 participants | 18 participants | 36 participants |

| | YES | 18 (100%) | 18 (100%) | 36 (100%) |
|---|---|---|---|---|
| Patent Ductus Arteriosus (PDA) at birth | | | | |
| Measure Type: Count of Participants | | | | |
| Unit of measure: Participants | | | | |
| | Number<br>Analyzed | 18 participants | 18 participants | 36 participants |
| | Present | 7 (38.9%) | 4 (22.2%) | 11 (30.6%) |

### **Outcome Measures**

### 1. Primary Outcome

| Title | Treatment failure |
|---|---|
| Description | hypoxia (FiO2 requirement >0.35), respiratory acidosis (pH < 7.2 & PCO 2 |
| | > 60 mm Hg) or major apnea requiring mask ventilation or >4 episodes/hour. |
| | Rescue treatment with NIPPV was also considered as treatment failure. |
| Time Frame | 72 hours |

#### **Outcome Measure Data**

### • Analysis Population Description

| Arm/Group Title | NI-NAVA | NIPPV |
|---|---|---|
| Arm/Group Description: | Non-invasive Neurally adjusted ventilatory assist (NAVA) after extubation in preterm infants | Non-invasive positive pressure ventilation (NIPPV) after extubation in preterm infants |
| Overall Number of<br>Participants Analyzed | 18 | 18 |
| Measure Type: Count of Participants | | |
| Unit of measure: Participants | | |
| | 1 (5.5%) | 0 (0%) |

| Statistical Analysis Overview | Comparison Group Selection | NI-NAVA, NIPPV |
|---|---|---|
| | Comments | [Not Specified] |
| | Type of Statistical Test | Superiority or Other |
| | Comments | [Not Specified] |
| Statistical Test of Hypothesis | P-Value | 0.310 |
| | Comments | [Not Specified] |
| | Method | Pearson's chi-square |
| | Comments | [Not Specified] |
| Method of Estimation | Estimation Parameter | |
| | Estimated Value | |
| | Confidence Interval | |
| | Parameter Dispersion | |
| | Estimation Comments | |

## 2. Primary Outcome

| Title | Reintubation |
|---|---|
| Description | Treatment failure leading to reintubation of infant within 72 hours |
| Time Frame | 72 hours |

## **Outcome Measure Data**

## • Analysis Population Description

The analysis was "per protocol". 36 patients who had completed the study was used for the analysis.

| Arm/Group Title | NI-NAVA | NIPPV |
|---|---|---|
| Arm/Group Description: | Non-invasive Neurally adjusted ventilatory assist (NAVA) after extubation in preterm infants | Non-invasive positive pressure ventilation (NIPPV) after extubation in preterm infants |
| Overall Number of<br>Participants Analyzed | 18 | 18 |
| Measure Type: Count of Participants | | |
| Unit of measure: Participants | | |
| | 4 (22.2%) | 2 (11.1%) |

| Statistical Analysis Overview | Comparison Group Selection | NI-NAVA, NIPPV |
|---|---|---|
| | Comments | [Not Specified] |
| | Type of Statistical Test | Superiority or Other |
| | Comments | [Not Specified] |
| Statistical Test of Hypothesis | P-Value | 0.371 |
| | Comments | [Not Specified] |
| | Method | Pearson's chi-square |
| | Comments | [Not Specified] |

| Method of Estimation | Estimation Parameter |
|----------------------|----------------------|
| | Estimated Value |
| | Confidence Interval |
| | Parameter Dispersion |
| | Estimation Comments |

| Title | Intraventricular Hemorrhage |
|---|---|
| Description | IVH (grades III & IV) classified according to Papile et al after evaluation of head ultrasound by a pediatric radiologist |
| Time Frame | 72 hours |

#### **Outcome Measure Data**

### • Analysis Population Description

| Arm/Group Title | NI-NAVA | NIPPV |
|---|---|---|
| Arm/Group Description: | Non-invasive Neurally adjusted | Non-invasive positive |
| | ventilatory assist (NAVA) after | pressure ventilation (NIPPV) |
| | extubation in preterm infants | after extubation in preterm |
| | | infants |
| Overall Number of | 18 | 18 |
| Participants Analyzed | | |

| Measure Type: Count of | | |
|-------------------------------|-----------|--------|
| Participants | | |
| Unit of measure: Participants | | |
| measure. Tarticipants | | |
| | 2 (11.1%) | 0 (0%) |

| Statistical Analysis Overview | Comparison Group Selection | NI-NAVA, NIPPV |
|---|---|---|
| | Comments | [Not Specified] |
| | Type of Statistical Test | Superiority or Other |
| | Comments | [Not Specified] |
| Statistical Test of Hypothesis | P-Value | 0.486 |
| | Comments | [Not Specified] |
| | Method | Fisher's exact |
| | Comments | [Not Specified] |
| Method of Estimation | Estimation Parameter | |
| | Estimated Value | |
| | Confidence Interval | |
| | Parameter Dispersion | |
| | Estimation Comments | |

# 4. Secondary Outcome

| Title | Necrotizing Enterocolitis |
|---|---|
| Description | Necrotizing enterocolitis defined according to modified Bell's criteria (stage 2 to 3) |
| Time Frame | 72 hours |

### **Outcome Measure Data**

## • Analysis Population Description

The analysis was "per protocol". 36 patients who had completed the study was used for the analysis.

| Arm/Group Title | NI-NAVA | NIPPV |
|---|---|---|
| Arm/Group Description: | Non-invasive Neurally adjusted ventilatory assist (NAVA) after | Non-invasive positive pressure ventilation (NIPPV) |
| | extubation in preterm infants | after extubation in preterm infants |
| Overall Number of<br>Participants Analyzed | 18 | 18 |
| Measure Type: Count of Participants | | |
| Unit of measure: Participants | | |
| | 4 (22.2%) | 0 (0%) |

| <b>Statistical Analysis Overview</b> | Comparison Group Selection | NI-NAVA, NIPPV |
|---|---|---|

| | Comments | [Not Specified] |
|---|---|---|
| | Type of Statistical Test | Superiority or Other |
| | Comments | [Not Specified] |
| <b>Statistical Test of Hypothesis</b> | P-Value | 0.034 |
| | Comments | [Not Specified] |
| | Method | Pearson's chi-square |
| | Comments | [Not Specified] |
| Method of Estimation | Estimation Parameter | |
| | Estimated Value | |
| | Confidence Interval | |
| | Parameter Dispersion | |
| | Estimation Comments | |

| Title | Pneumothorax |
|-------------|---------------------------------------------------------|
| Description | Air leak within pleural cavity diagnosed radiologically |
| Time Frame | 72 hours |

#### **Outcome Measure Data**

## • Analysis Population Description

| Arm/Group Title | NI-NAVA | NIPPV |
|---|---|---|
| Arm/Group Description: | Non-invasive Neurally adjusted ventilatory assist (NAVA) after extubation in preterm infants | Non-invasive positive pressure ventilation (NIPPV) after extubation in preterm infants |
| Overall Number of<br>Participants Analyzed | 18 | 18 |
| Measure Type: Count of Participants | | |
| Unit of measure: Participants | | |
| | 0 (0%) | 0 (0%) |

| Statistical Analysis Overview | Comparison Group Selection | NI-NAVA, NIPPV |
|---|---|---|
| | Comments | [Not Specified] |
| | Type of Statistical Test | Superiority or Other |
| | Comments | [Not Specified] |
| <b>Statistical Test of Hypothesis</b> | P-Value | - |
| | Comments | [Not Specified] |
| | Method | - |
| | Comments | [Not Specified] |
| Method of Estimation | Estimation Parameter | |
| | Estimated Value | |

| Confidence Interval |
|----------------------|
| Parameter Dispersion |
| Estimation Comments |

| Title | GI Perforation |
|---|---|
| Description | Gastrointestinal perforation diagnosed radiologically or at operation |
| Time Frame | 72 hours |

#### **Outcome Measure Data**

## • Analysis Population Description

| Arm/Group Title | NI-NAVA | NIPPV |
|---|---|---|
| Arm/Group Description: | Non-invasive Neurally adjusted ventilatory assist (NAVA) after extubation in preterm infants | Non-invasive positive pressure ventilation (NIPPV) after extubation in preterm infants |
| Overall Number of<br>Participants Analyzed | 18 | 18 |
| Measure Type: Count of Participants Unit of | | |
| measure: Participants | | |

| 1 (5.6%) | 0 (0%) |
|----------|--------|

| Statistical Analysis Overview | Comparison Group Selection | NI-NAVA, NIPPV |
|---|---|---|
| | Comments | [Not Specified] |
| | Type of Statistical Test | Superiority or Other |
| | Comments | [Not Specified] |
| Statistical Test of Hypothesis | P-Value | 0.310 |
| | Comments | [Not Specified] |
| | Method | Pearson's chi-square |
| | Comments | [Not Specified] |
| Method of Estimation | Estimation Parameter | |
| | Estimated Value | |
| | Confidence Interval | |
| | Parameter Dispersion | |
| | Estimation Comments | |

## 7. Secondary Outcome

| Title | Sepsis |
|---|---|
| Description | Nosocomial sepsis defined as presence of clinical signs of sepsis or positive blood or cerebrospinal fluid (CSF) cultures taken after five days of age |
| Time Frame | 72 hours |

#### **Outcome Measure Data**

### • Analysis Population Description

The analysis was "per protocol". 36 patients who had completed the study was used for the analysis.

| Arm/Group Title | NI-NAVA | NIPPV |
|---|---|---|
| Arm/Group Description: | Non-invasive Neurally adjusted ventilatory assist (NAVA) after extubation in preterm infants | Non-invasive positive pressure ventilation (NIPPV) after extubation in preterm |
| | 1 | infants |
| Overall Number of | 18 | 18 |
| Participants Analyzed | | |
| Measure Type: Count of Participants | | |
| Unit of measure: Participants | | |
| | 2 (11.1%) | 2 (11.1%) |

| Statistical Analysis Overview | Comparison Group Selection | NI-NAVA, NIPPV |
|---|---|---|
| | Comments | [Not Specified] |
| | Type of Statistical Test | Superiority or Other |
| | Comments | [Not Specified] |
| Statistical Test of Hypothesis | P-Value | 1.000 |

| | Comments | [Not Specified] |
|----------------------|----------------------|----------------------|
| | Method | Pearson's chi-square |
| | Comments | [Not Specified] |
| Method of Estimation | Estimation Parameter | |
| | Estimated Value | |
| | Confidence Interval | |
| | Parameter Dispersion | |
| | Estimation Comments | |

| Title | Retinopathy of prematurity |
|---|---|
| Description | Retinopathy of prematurity (ROP) stage 3 or greater according to International classification |
| Time Frame | 72 hours |

#### **Outcome Measure Data**

## • Analysis Population Description

| Arm/Group Title | NI-NAVA | NIPPV |
|---|---|---|
| Arm/Group Description: | Non-invasive Neurally adjusted | Non-invasive positive |
| | ventilatory assist (NAVA) after | pressure ventilation (NIPPV) |
| | extubation in preterm infants | |

| | | after extubation in preterm |
|------------------------|-----------|-----------------------------|
| | | infants |
| Overall Number of | 18 | 18 |
| Participants Analyzed | | |
| Measure Type: Count of | | |
| Participants | | |
| Unit of | | |
| measure: Participants | | |
| | 2 (11.1%) | 1 (5.6%) |

| Statistical Analysis Overview | Comparison Group Selection | NI-NAVA, NIPPV |
|---|---|---|
| | Comments | [Not Specified] |
| | Type of Statistical Test | Superiority or Other |
| | Comments | [Not Specified] |
| <b>Statistical Test of Hypothesis</b> | P-Value | 0.546 |
| | Comments | [Not Specified] |
| | Method | Pearson's chi-square |
| | Comments | [Not Specified] |
| Method of Estimation | Estimation Parameter | |
| | Estimated Value | |
| | Confidence Interval | |
| | Parameter Dispersion | |

| Estimation Comments |
|---------------------|

## **Adverse Events**

| Time Frame | 72 hours | |
|---|---|---|
| Adverse Event | [Not Specified] | |
| Reporting | | |
| Description | | |
| | <u> </u> | |
| Arm/Group Title | NI-NAVA | NIPPV |
| Arm/Group | Non-invasive Neurally adjusted | Non-invasive positive pressure |
| Description | ventilatory assist (NAVA) after | ventilation (NIPPV) after extubation |
| | extubation in preterm infants | in preterm infants |
| All-Cause Mortality | | |
| | NI-NAVA | NIPPV |
| | Affected / at Risk (%) | Affected / at Risk (%) |
| Total | 2/18 (11.1%) | 1/18 (5.6%) |
| Serious Adverse Event | s | |
| | NI-NAVA | NIPPV |
| | Affected / at Risk (%) | Affected / at Risk (%) |
| Total | 0/18 (0.00%) | 0/18 (0.00%) |
| <b>▼</b> Other (Not Includin | g Serious) Adverse Events | |
| Frequency Threshold | 5% | |
| for Reporting Other | | |
| Adverse Events | | |
| | NI-NAVA | NIPPV |
| | Affected / at Risk (%) | Affected / at Risk (%) |

| Total | 0/18 (0.00%) | 0/18 (0.00%) |
|-------|--------------|--------------|